CLINICAL TRIAL: NCT02417766
Title: NIAID Clinical Center Genomics Opportunity Protocol
Status: Completed | Type: Observational
Sponsor: National Institute of Allergy and Infectious Diseases (NIAID) (NIH)
Responsible Party: Sponsor
Organization: National Institutes of Health Clinical Center (CC) (NIH)
Other Study IDs: 150113; 15-I-0113
Record Dates: First submitted 2015-04-15; First posted 2015-04-16 (Estimated); Last update posted 2023-03-16 (Actual); Status verified 2023-03

CONDITIONS: Immune Disorders
Keywords: Genetic Testing; Secondary Findings; Immune-Mediated Disorders; Whole Exome Sequencing; Natural History
MeSH Terms: conditions — Immune System Diseases

STUDY DESIGN:
Observational Model: Family Based | Time Perspective: Prospective
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (2):
- Family Members: Family members to the patients
- Patient: Patients here at NIH

SUMMARY:
Background:

- There are many types of immune disorders. These range from rare immune deficiencies to allergies to autoimmune disease like rheumatoid arthritis. Genes are the instructions our body uses to work and develop. A new technology called whole exome sequencing may help find the cause of these disorders. Whole exome sequencing is a way to look at many genes at once for errors. Researchers hope to find new gene changes that lead to immune disorders. Additionally, researchers are interested in finding the best way to manage unexpected but important findings by whole exome sequencing.

Objectives:

- To better understand genetic causes of immune system disorders. Also, to better understand people s thoughts and feelings about immune system disorders and new genomic testing.

Eligibility:

- People ages 0 100 with an immune disorder or a relative with an immune disorder. People must be at least 2 to be evaluated at the NIH clinical center. People must be at least 12 to do the survey/interview portion of the study.

Design:

* Participants will have their genes sequenced. They may be asked for a new sample of blood.
* If participants cannot come for a study visit, they can have a blood sample collected by their local lab or doctor and sent by mail.
* Researchers may or may not find the cause of the participant s immune disorder. Participants will learn that information. Some participants may be asked to return to NIH to get results and have more tests.
* Researchers may share information with other studies. The data will be anonymous.
* For the survey part of the study, participants will answer questions about their or their relative s immune disorder. They will also answer about their thoughts and feelings about genomic testing.
* Some participants will be asked for a brief interview to ask more about the survey topics. There may be more follow-up after several months.

DETAILED DESCRIPTION:
Investigators at National Institute of Allergy and Infectious Diseases (NIAID) are actively developing the infrastructure and capability for identifying the cause of heterogeneous immune-mediated disorders through whole exome and whole genome sequencing (WES/WGS). This effort received additional support through the establishment of the NIAID Clinical Genomics Program (CGP), a Division of Intramural Research (DIR)-supported cross-lab collaboration to increase the effectiveness of NIAID s basic and applied genomic research. The disorders under investigation include primary immunodeficiencies, immune homeostasis disorders, autoimmune conditions, and allergic diseases for which the hypothesized causative genetic mutations(s) have not yet been identified. Given recent discoveries of the genetic bases of many immunological disorders, we are also expanding the disorders studied to include those with prominent extra-immune manifestations in which a strong inherited immunological pathogenic basis has been identified; such as the Pediatric Autoimmune Neuropsychiatric Disorders associated with Streptococcal infections (PANDAS) or Sydenham s chorea. Despite the breadth of clinical presentations under investigation, these immune-mediated disorders share significant overlap in underlying molecular pathophysiology and thus represent a coherent study target.

This protocol will facilitate the discovery of genes contributing to selected immune-mediated disorders as well as generating experience with genetic secondary finding disclosure and will further assess participant s perceptions and preference for WES and future secondary finding procedures. Ultimately, a better understanding of the genetic contribution to immune dysregulation will not only provide valuable diagnostic and, potentially, prognostic information to affected families, but also has the potential to lead to the development of novel therapeutic targets. Further, developing experience-tested and evidenced-based procedures for secondary finding management is beneficial for NIAID CGP researchers and participants.

This protocol is specific for genetic testing. Probands, or the affected person serving as the starting point for the genetic study of family, will be required to be enrolled on a primary protocol, which will execute the clinical and research evaluations. Unaffected relatives may be enrolled on this protocol only. Participants unable to travel to National Institutes of Health (NIH) Clinical Center (NIHCC) may be evaluated through mailin blood samples, although evaluation at the NIHCC is strongly preferred, particularly for affected participants. This study aims to enroll 200 participants for exome sequencing, including both patients and relatives with heterogeneous immune-mediate disorders; all participants receiving exome sequencing plus those who decline will be offered participation in the survey (i.e., up to the accrual ceiling of 200).

ELIGIBILITY:
* INCLUSION CRITERIA:

Whole Exome Sequencing with Secondary Findings Disclosure

The following inclusion criteria apply to all research participants on this protocol:

1. Age 0-100 years old. Clinical evaluation at the NIHCC requires age >2 years. Affected relatives <2 years of age may be included in genetic family studies despite the fact that he/she is too young for evaluation at the clinical center. Including affected relatives in family-based whole exome sequencing is critically important, even if the study team has to rely only on medical records because NIHCC evaluation is not permitted due to age.
2. Willingness to allow sharing of genetic information in shared controlled access databases like dbGaP.
3. Willingness to receive secondary finding report.

Probands (i.e., affected individuals serving as the starting point for genetic study of a family) must have:

1. Primary enrollment on a NIH Institutional Review Board (IRB) approved protocol (e.g., 05-I-0213 or 93-I-0063), which will execute the majority of clinical and research evaluations.
2. A suspected genetic basis for the presenting immune disorder with features including but not limited to autoimmunity, autoinflammatory conditions, lymphadenopathy, end-organ dysfunction, unusual infections, allergies, or laboratory abnormalities consistent with immune dysregulation that has not been previously identified and/or with a family history suggesting genetically-based immune dysfunction (e.g., similar phenotypes among relatives and/or consanguinity).

EXCLUSION CRITERIA:

Any participant can be excluded for the following:

1. Any condition which in the opinion of the investigator may interfere with the research that is the focus of this protocol.

Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Study Population: NIAID Investigators and NIMH -PANDAS patients
Sampling Method: Non-Probability Sample
Enrollment: 139 (Actual)
Dates: Start 2015-06-29 (Actual); Primary Completion 2019-01-22 (Actual); Study Completion 2019-01-22 (Actual)

PRIMARY OUTCOMES:
To discover genes contributing to selected immunemediated disorders | 6 - 8 months after blood analysis
  determination of discrete genotypephenotype association for selected immune-mediated disorders

SECONDARY OUTCOMES:
Secondary Findings -To generate experience with secondary finding disclosure among NIAID genomic researchers and further assess the perceptions and preferences among NIAID study participants for WES including secondary finding analysis and discl... | 6 - 8 months after blood analysis
  to better understand participants WES-related perceptions and preferences, including secondary finding analysis and disclosure in order to inform future practice.

CONTACTS AND LOCATIONS:
Overall Officials: Morgan N Similuk, Principal Investigator — National Institute of Allergy and Infectious Diseases (NIAID)
Locations (1):
- National Institutes of Health Clinical Center, Bethesda, Maryland, United States

REFERENCES:
- [Background] Similuk MN, Yan J, Setzer MR, Jamal L, Littel P, Lenardo M, Su HC. Exome sequencing study in a clinical research setting finds general acceptance of study returning secondary genomic findings with little decisional conflict. J Genet Couns. 2021 Jun;30(3):766-773. doi: 10.1002/jgc4.1367. Epub 2020 Dec 15. PMID 33320394
- See also: NIH Clinical Center Detailed Web Page — https://clinicalstudies.info.nih.gov/cgi/detail.cgi?B_2015-I-0113.html